CLINICAL TRIAL: NCT03298061
Title: Mepolizumab Long-term Access Programme for Subjects Who Participated in Study MEA115921 (Placebo-controlled Study of Mepolizumab in the Treatment of Eosinophilic Granulomatosis With Polyangiitis in Subjects Receiving Standard-of-care Therapy)
Brief Title: Long-term Access Program (LAP) of Mepolizumab for Subjects Who Participated in Study MEA115921
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116841; 2014-003162-25 (EudraCT Number)
Expanded Access: NCT00244686 (No longer available)
Record Dates: First submitted 2017-09-27; First posted 2017-09-29 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Churg-Strauss Syndrome; Eosinophilic Granulomatosis With Polyangiitis
Keywords: Eosinophilic Granulomatosis; MEA115921; Polyangiitis; Long-term access program; mepolizumab
MeSH Terms: conditions — Churg-Strauss Syndrome; Systemic Vasculitis | interventions — mepolizumab; Prednisolone

STUDY DESIGN:
Intervention Model Description: Subjects who participated in clinical study MEA115921 and require a dose of prednisolone (or equivalent) of >=5 mg/day for adequate control of their EGPA will be included in this study based on the confirmation of their eligibility by GSK Medical Monitor. Eligible subjects will receive subcutaneously administered mepolizumab at a dose of 300 mg SC every 4 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects from clinical study MEA115921 (Experimental): Subjects who participated in clinical study MEA115921 and who require a dose of prednisolone (or equivalent) of 5 mg/day for adequate control of their EGPA will be included. Eligible subjects will receive subcutaneously administered mepolizumab at a dose of 300 mg SC every 4 weeks.
  Interventions: Drug: Mepolizumab; Drug: Prednisolone

INTERVENTIONS:
Drug: Mepolizumab — Mepolizumab will be available as lyophilized powder for injection to be reconstituted with sterile water for injection, prior to use. Subjects will be dosed with mepolizumab at a dose of 300 mg which will be administered as three separate 100 mg SC injections every 4 weeks. The injections will be administered into any of the upper arm, thigh or anterior abdominal wall.
Drug: Prednisolone — Subjects who require a dose of prednisolone (or equivalent) of 5 mg/day for adequate control of their EGPA will be included.

SUMMARY:
Eosinophilic Granulomatosis with Polyangiitis (EGPA), also referred to as Churg-Strauss syndrome, is a rare hyper-eosinophilic syndrome. Eosinophilia is central to the pathophysiology of EGPA and interleukin-5 (IL-5) is a key cytokine regulating the life-cycle of the eosinophil. Neutralization of IL-5 with mepolizumab, an anti-IL5 monoclonal antibody, therefore offers a potential therapeutic option for EGPA. The objective of study MEA115921 was to investigate the efficacy and safety of mepolizumab compared with placebo wherein the subjects were randomized to receive either: 300 milligram (mg) mepolizumab or Placebo subcutaneous (SC) injection every 4 weeks in addition to their background standard-of-care therapy. Subjects were treated for a period of 52 weeks and then followed up for a further 8 weeks to study completion at Week 60. This is a LAP to support provision of open-label mepolizumab on an individual basis to eligible subjects who participated in clinical study MEA115921 and who require a dose of prednisolone (or equivalent) of >=5 milligrams per day (mg/day) for adequate control of their EGPA. Eligible subjects can initiate mepolizumab under this LAP within a 6-month period starting from completion of study MEA115921 (that is, at Week 60) or, in case of premature discontinuation from study MEA115921, the subjects will initiate mepolizumab at the time point that would have been Week 60 if the subject had completed the study. Eligible subjects will receive subcutaneously administered mepolizumab at a dose of 300 mg SC every 4 weeks. Eligible subjects will continue to receive mepolizumab under this LAP until mepolizumab is commercially licensed for the treatment of EGPA in the relevant country or until GlaxoSmithKline (GSK) discontinues the program or until the subject meets any of the withdrawal/stopping criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subject participated in study MEA115921.
* Subject has either: a) completed study MEA115921 to Week 60, that is, completion of follow up period, or b) if the subject was withdrawn prematurely from study MEA115921, the subject has reached the date of what would have been the Week 60 if the subject had completed the study, that is, 60 weeks from Baseline (Visit 2).
* At or up to 6 months after the MEA115921 Week 60 time- point the subject requires a dose of prednisolone (or equivalent) of >=5 mg/day for adequate control of their EGPA.
* The treating physician requesting mepolizumab under this LAP considers the benefits of treatment with mepolizumab outweigh the risks for the individual subject.
* To be eligible for mepolizumab treatment under this LAP, females of childbearing potential (FCBP) must commit to consistent and correct use of an acceptable method of birth control, beginning with consent, for the duration of the treatment with mepolizumab and for 4 months after the last mepolizumab administration.
* The subject consents to receiving treatment with mepolizumab under this LAP.

Exclusion Criteria:

* A current malignancy or history of cancer in remission for less than 12 months (Subjects who had localized carcinoma (that is, basal or squamous cell) of the skin which was resected for cure will not be excluded).
* Subject has other clinically significant medical conditions uncontrolled with standard of care therapy not associated with EGPA, example, unstable liver disease, uncontrolled cardiovascular disease, ongoing active infectious disease requiring systemic treatment.
* Subject is pregnant or breastfeeding. Subjects should not be considered for continued treatment if they plan to become pregnant during the course of treatment with mepolizumab.
* Subject has a known allergy or intolerance to a monoclonal antibody or biologic therapy including mepolizumab.
* Subject had an adverse event (serious or non-serious) considered related to study treatment whilst participating in study MEA115921 which resulted in permanent withdrawal of study treatment.
* Subject is receiving treatment with another biological therapy such as a monoclonal antibody therapy or intravenous (IV) immunoglobulin therapy without prior agreement from the GSK Medical Monitor.
* Subjects who have received treatment with an investigational drug within the past 30 days or 5 terminal phase half-lives of the drug whichever is longer, prior to initiation of mepolizumab treatment under this LAP (this also includes investigational formulations of marketed products).
* Subject is currently participating in any other interventional clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (31):
- United States (13):
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Mempis, Tennessee
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, St. George, Utah
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Bellevue, Washington
- GSK Investigational Site, Brussels, Belgium
- GSK Investigational Site, Hamilton, Ontario, Canada
- France (6):
  - GSK Investigational Site, Bron
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Priest-en-Jarez
  - GSK Investigational Site, Suresnes
- Germany (5):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Kirchheim -Teck, Baden-Wurttemberg
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Bad Bramstedt, Schleswig-Holstein
  - GSK Investigational Site, Jena, Thuringia
- Japan (2):
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Miyagi
- United Kingdom (3):
  - GSK Investigational Site, Portsmouth, Hampshire
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Leicester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who participated in clinical study MEA115921 and required a dose of prednisolone (or equivalent) of greater than or equal to (>=) 5 milligrams per day (mg/day) for adequate control of their Eosinophilic Granulomatosis with Polyangiitis (EGPA) were included in this study based on their eligibility. Eligible participants received subcutaneous (SC) injection of mepolizumab 300 milligrams (mg) every 4 weeks.
Pre-assignment Details: A total of 100 participants entered the study and received mepolizumab.
Groups:
- Mepolizumab 300 mg: Participants who participated in clinical study MEA115921, who required additional dose of >=5 milligrams per day (mg/day) prednisolone for adequate control of their Eosinophilic Granulomatosis with Polyangiitis (EGPA) received 300 milligrams (mg) mepolizumab subcutaneous (SC) injection every 4 weeks.
Period: Overall Study
Arm/Group | Mepolizumab 300 mg
Started | 100
Completed | 73
Not Completed | 27
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 6
Not completed — Protocol Violation | 1
Not completed — Physician Decision | 7
Not completed — Withdrawal by Subject | 10

BASELINE CHARACTERISTICS:
Arm/Group | Mepolizumab 300 mg
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 49.6 (13.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 1
  ASIAN - JAPANESE HERITAGE | 6
  ASIAN - SOUTH EAST ASIAN HERITAGE | 2
  WHITE - ARABIC/NORTH AFRICAN HERITAGE | 1
  WHITE - WHITE/CAUCASIAN/EUROPEAN HERITAGE | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; other important medical events based on medical or scientific judgment; and is associated with liver injury and impaired liver function. Additionally, systemic (that is, allergic/hypersensitivity and non-allergic) reactions and local injection site reactions were recorded throughout the treatment and follow-up period.
Time Frame: Up to approximately 89 Months
Population: Safety Population consisted of all participants who received at least one dose of open label mepolizumab. On-treatment AEs and on-treatment SAEs are the events occurring on/after the first dose of open-label mepolizumab date and before/on last dose of mepolizumab + 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 300 mg
Number analyzed (Participants) | 100
Participants
  AE | 98
  SAE | 38

ADVERSE EVENTS:
Time Frame: Up to approximately 89 Months
Description: Adverse events (AEs) and Serious adverse event (SAEs) were collected for all participants within the safety population which comprised of all participants who received at least one dose of open-label mepolizumab.
Arm/Group | Mepolizumab 300 mg
All-Cause Mortality (participants affected / at risk) | 1/100
Serious Adverse Events (participants affected / at risk) | 38/100
Other Adverse Events (participants affected / at risk) | 97/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab 300 mg (N=100)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (2)
Myocardial infarction (Cardiac disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (2)
Rectal ulcer (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Eosinophilic granulomatosis with polyangiitis (Immune system disorders) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2)
Bursitis infective (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Chronic sinusitis (Infections and infestations) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Hepatitis E (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (4)
Pneumonia (Infections and infestations) | 3 (7)
Pneumonia pneumococcal (Infections and infestations) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Salpingitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cervical cord compression (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Stress (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (2)
Renal colic (Renal and urinary disorders) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vocal cord dysfunction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab 300 mg (N=100)
Anaemia (Blood and lymphatic system disorders) | 4 (5)
Cataract (Eye disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 6 (8)
Abdominal pain upper (Gastrointestinal disorders) | 4 (26)
Diarrhoea (Gastrointestinal disorders) | 14 (16)
Gastritis (Gastrointestinal disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 14 (18)
Vomiting (Gastrointestinal disorders) | 10 (10)
Asthenia (General disorders) | 3 (4)
Fatigue (General disorders) | 10 (12)
Influenza like illness (General disorders) | 6 (8)
Injection site haematoma (General disorders) | 4 (5)
Injection site reaction (General disorders) | 13 (29)
Oedema peripheral (General disorders) | 3 (3)
Pyrexia (General disorders) | 7 (14)
Eosinophilic granulomatosis with polyangiitis (Immune system disorders) | 4 (4)
Acute sinusitis (Infections and infestations) | 8 (14)
Bronchitis (Infections and infestations) | 29 (47)
COVID-19 (Infections and infestations) | 6 (7)
Conjunctivitis (Infections and infestations) | 3 (4)
Cystitis (Infections and infestations) | 3 (4)
Ear infection (Infections and infestations) | 8 (9)
Gastroenteritis (Infections and infestations) | 8 (11)
Herpes simplex (Infections and infestations) | 4 (4)
Influenza (Infections and infestations) | 10 (12)
Lower respiratory tract infection (Infections and infestations) | 7 (21)
Nasopharyngitis (Infections and infestations) | 33 (113)
Oral candidiasis (Infections and infestations) | 5 (5)
Otitis media (Infections and infestations) | 4 (9)
Pharyngitis (Infections and infestations) | 4 (4)
Pneumonia (Infections and infestations) | 3 (3)
Pulpitis dental (Infections and infestations) | 3 (5)
Respiratory tract infection (Infections and infestations) | 13 (15)
Rhinitis (Infections and infestations) | 3 (6)
Sinusitis (Infections and infestations) | 30 (52)
Tooth abscess (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 31 (43)
Urinary tract infection (Infections and infestations) | 13 (16)
Viral infection (Infections and infestations) | 7 (8)
Viral upper respiratory tract infection (Infections and infestations) | 8 (8)
Arthropod bite (Injury, poisoning and procedural complications) | 5 (5)
Bone contusion (Injury, poisoning and procedural complications) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 8 (10)
Foot fracture (Injury, poisoning and procedural complications) | 5 (7)
Hand fracture (Injury, poisoning and procedural complications) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3)
Muscle strain (Injury, poisoning and procedural complications) | 4 (6)
Rib fracture (Injury, poisoning and procedural complications) | 6 (6)
Weight decreased (Investigations) | 5 (5)
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (29)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (19)
Bursitis (Musculoskeletal and connective tissue disorders) | 4 (4)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (18)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (13)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Dizziness (Nervous system disorders) | 8 (8)
Headache (Nervous system disorders) | 14 (42)
Hypoaesthesia (Nervous system disorders) | 3 (3)
Migraine (Nervous system disorders) | 3 (3)
Paraesthesia (Nervous system disorders) | 8 (8)
Sciatica (Nervous system disorders) | 4 (6)
Depression (Psychiatric disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 7 (8)
Dysuria (Renal and urinary disorders) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 26 (87)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 3 (17)
Rash (Skin and subcutaneous tissue disorders) | 15 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT03298061/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT03298061/SAP_001.pdf